CLINICAL TRIAL: NCT02597712
Title: Randomized, Placebo-controlled Trial of YF476, a Gastrin Receptor Antagonist, in Barrett's Esophagus
Brief Title: YF476 in Barrett's Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trio Medicines Ltd. (Industry)
Collaborators: Columbia University (Other); University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T-016
Record Dates: First submitted 2015-06-03; First posted 2015-11-05 (Estimated); Results first posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Barrett's Esophagus
Keywords: acid reflux; intragastric pH; gastrin; hypergastrinemia
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux | interventions — YF 476

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Patients will take 25 mg YF476 once daily for 12 weeks
  Interventions: Drug: YF476
- YF476 Placebo (Placebo Comparator): Patients will take matching placebo once daily for 12 weeks
  Interventions: Drug: YF476 placebo

INTERVENTIONS:
Drug: YF476 — gastrin receptor antagonist
  Other Names: netazepide
  Arms: Treatment
Drug: YF476 placebo — placebo
  Other Names: netazepide placebo
  Arms: YF476 Placebo

SUMMARY:
A phase 2, randomised, double-blind, out-patient trial to determine if YF476 is a safe and effective treatment in patients with Barrett's esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years, with histologically confirmed diagnosis of Barrett's esophagus (BE) without dysplasia. A prior endoscopy with biopsies read as indefinite for dysplasia is permitted if biopsies from the most recent endoscopy prior to study entry demonstrated BE without dysplasia.
* Minimum of 1 cm circumferential Barrett's mucosa on endoscopy or at least 2 cm maximal contiguous extent of Barrett's mucosa, as measured from the top of the gastric folds to the squamocolumnar junction (Prague criteria C>1, any M or any C, M>2).
* Proton pump inhibitor use at least once daily, for at least 12 months prior to enrolment, and stable dose of PPI for the 3 months before enrolment. Any PPI, dose, and frequency allowable.
* ECOG performance status <2 and Karnofsky >60%
* Normal organ and marrow function, defined as white blood cells >3 x 10e9, absolute neutrophil count >1.5 x 10e9, platelets >100 x 10e9, creatinine <1.5 mg/dL, total bilirubin <1.5 mg/dL, AST <100 U/L, ALT <100 U/L.
* Use of adequate contraception during the study, as follows;
* Post-menopausal women must have had their last menstrual period at least 1 year ago.
* Pre-menopausal women, who are sexually-active, must have had a hysterectomy or bilateral oophorectomy; or must use an intrauterine device (IUD), or spermicide with a diaphragm, cap or condom. Streroid contraceptives such as 'the pill' are not allowed unless in combination with one of the aforementioned barrier contraceptive methods.
* Men must use a condom and spermicide.
* Willingness to comply with all treatment and follow-up procedures.
* Ability to understand and the willingness to sign a written informed consent document.
* Up to date with all age-appropriate cancer screening tests, as per American Cancer Society guidelines, (Columbia University only), and no cancer screening tests planned for the next 21 weeks.

Exclusion Criteria:

* Histologically confirmed BE with high-grade dysplasia.
* Histologically confirmed diagnosis of invasive carcinoma of the esophagus.
* Histologically confirmed BE with low-grade dysplasia that has been diagnosed by at least 2 expert gastrointestinal pathologists.
* Prior endoscopic therapy for BE.
* Any history of esophageal or gastric surgery.
* History of atrophic gastritis, pernicious anemia, or Zollinger-Ellison syndrome.
* Participation in a trial of an IMP within the previous 28 days.
* Prolonged QTc interval >450 msec.
* History of allergic reactions attributed to compounds of similar chemical composition of YF476.
* History of baseline findings of:
* diabetes mellitus requiring insulin therapy
* pancreatitis (baseline amylase and/or lipase >2.0 x ULN)
* hepatitis B, hepatitis C or HIV
* malabsorption syndrome or inability to swallow or retain oral medicine
* major surgery <28 days prior to enrolment
* ECOG performance status >2
* another cancer within 3 years except for basal carcinoma of the skin or cervical carcinoma in-situ
* also, any clinically significant and uncontrolled major morbidity including but not limited to: serious cardiac disease (unstable angina, s/p myocardial infarction <1 month); respiratory disease (advanced COPD or pulmonary fibrosis); uncontrolled hypertension; active systemic infection; or psychiatric illness/social situations that would limit compliance with study requirements.
* Certain medicines and herbal remedies taken during the 7 days before the start of the study drug.
* A history of cancer >3 years from the time of enrolment, and the patient is not up to date with surveillance for that cancer (based on the American Cancer Society guidelines, Columbia University only), has evidence of cancer at the time of enrolment, or has surveillance tests planned within 21 weeks after enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-05-15 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian A Abrams, MD MS, Principal Investigator — Columbia University
Locations (2):
- Columbia University, Division of Digestive & Liver Diseases, New York, New York, United States
- MRC Cancer Unit, University of Cambridge, Cambridge, Cambridgeshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three patients were enrolled but failed screening due to elevated lipase, prolonged QTc or being diagnosed with lymphoma.
Period: Overall Study
Arm/Group | Treatment | YF476 Placebo
Started | 13 | 11
Completed | 10 | 10
Not Completed | 3 | 1
Not completed — Baseline biopsies showed indefinite for dysplasia | 2 | 0
Not completed — Baseline biopsies showed low grade dysplasia | 1 | 0
Not completed — Recurrent metastatic prostate cancer | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | YF476 Placebo | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12
  United Kingdom | 6 | 6 | 12
Ki67 expression [Mean (Standard Deviation); unit: cells/mm^2] | 1539 (514) | 1556 (622) | 1548 (559)
Fasting serum gastrin concentration (marker of gastric acid suppression) [Mean (Standard Deviation); unit: pmol/L] | 66.74 (41.736) | 51.85 (29.104) | 56.45 (35.997)
Fasting plasma CgA concentration (marker of ECL cell hyperplasia) [Mean (Standard Deviation); unit: nmol/L] | 12.93 (17.210) | 9.12 (4.98) | 11.18 (13.00)

OUTCOME MEASURES:

1. Primary Outcome: Change in Ki67 Biomarker Expression
Description: Esophagogastroduodenoscopy (EGD) was performed to enable taking biopsies for assessment of Ki67 expression, a marker of cellular proliferation. Ki67 expression was assessed by immunohistochemistry and calculating the number of Ki67 positive cells per mm^2 of Barrett's epithelium.
Time Frame: Baseline and Week 12
Population: 3 patients in the treatment arm and 1 patient in the placebo arm were withdrawn from the study due to reasons unrelated to the treatment. Therefore, Week 12 data show results from 10 patients per arm.
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | Treatment | YF476 Placebo
Number analyzed (Participants) | 13 | 11
cells/mm^2
  Baseline | 1539 (514) | 1556 (622)
  Week 12: number analyzed (Participants) | 10 | 10
  Week 12 | 1575 (620.7) | 1864 (640.3)

2. Secondary Outcome: Expression of Biomarkers Potentially Associated With Esophageal Adenocarcinoma (EAC)
Description: Blood samples were taken for assay of biomarkers associated with esophageal adenocarcinoma. Changes in biomarker expression were derived from RNA-Sequencing and calculated as log-fold change comparing the treatment group to the placebo group. The nature of how results are derived by RNA-sequencing means summary statistics cannot be generated individually for each arm and a value has not been calculated for each individual participant. Therefore, results are reported as the relative change in biomarker expression in the treatment arm compared to the placebo arm.
Time Frame: Week 12
Population: 3 patients in the treatment arm were withdrawn from the study due to reasons unrelated to the treatment. Therefore, results are reported for 10 patients.
Measure: Number; unit: relative log-fold change
Arm/Group | Treatment
Number analyzed (Participants) | 10
relative log-fold change
  CCK2R, Week 12 | -1.19
  PTGS2, Week 12 | 0.31
  DCLK1, Week 12 | -0.34

3. Secondary Outcome: Abundance of Biomarkers of Gastric Acid Suppression
Description: Blood samples were taken to assess the effects of YF476 on fasting serum gastrin, a marker of gastric acid suppression
Time Frame: Week 4, Week 6, Week 8, Week 12 and Follow-up (4 weeks after stopping YF476 treatment)
Population: After 6 patients (3 per treatment) had their Week 4 and 8 visits, the protocol was amended so that those visits were replaced by a single visit at Week 6 in order to reduce the total number of visits.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Treatment | YF476 Placebo
Number analyzed (Participants) | 10 | 10
pmol/L
  Week 4: number analyzed (Participants) | 3 | 3
  Week 4 | 242.6 (142.3) | 43.6 (9.9)
  Week 6: number analyzed (Participants) | 7 | 8
  Week 6 | 103.3 (89.9) | 63.9 (32.2)
  Week 8: number analyzed (Participants) | 3 | 3
  Week 8 | 234.3 (156.5) | 96.4 (54.2)
  Week 12 | 146.8 (112.8) | 49.2 (20.4)
  Follow-up | 94.9 (78.8) | 64.7 (37.7)

4. Secondary Outcome: Abundance of Biomarkers of ECL Cell Hyperplasia
Description: Blood samples were taken to assess the effects of YF476 on fasting plasma CgA, a marker of ECL cell hyperplasia
Time Frame: Week 4, Week 6, Week 8, Week 12 and Follow-up (4 weeks after stopping YF476 treatment)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Treatment | YF476 Placebo
Number analyzed (Participants) | 10 | 10
nmol/L
  Week 4: number analyzed (Participants) | 3 | 3
  Week 4 | 3.9 (1.8) | 8.8 (3.7)
  Week 6: number analyzed (Participants) | 7 | 8
  Week 6 | 1.8 (0.9) | 16.9 (9.8)
  Week 8: number analyzed (Participants) | 3 | 3
  Week 8 | 3.8 (1.8) | 10.9 (6.0)
  Week 12 | 2.9 (2.5) | 10.6 (7.4)
  Follow-up | 19.8 (26.1) | 11.9 (7.2)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Any untoward medical occurrence in a study participant that does not necessarily have a causal relationship with the treatment
Arm/Group | Treatment | YF476 Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/11
Other Adverse Events (participants affected / at risk) | 13/13 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=13) | YF476 Placebo (N=11)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=13) | YF476 Placebo (N=11)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal upper pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gatrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulveration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhintis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT02597712/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT02597712/SAP_001.pdf